CLINICAL TRIAL: NCT03330678
Title: Change in Human Gut Flora and in Immune Functions Following Probiotic Administration
Brief Title: Effect of Probiotic Administration on Gut Flora Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Rakesh Aggarwal, Professor, Gastroenterology, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-70-EMP-61
Record Dates: First submitted 2017-10-26; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Probiotics
Keywords: Probiotic; Gut microbiome; VSL#3
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Healthy young women will be given VSL#3 for 4 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Probiotic (VSL#3) (Experimental): Probiotics will be given to women included in study arm
  Interventions: Dietary Supplement: Probiotic (VSL#3)

INTERVENTIONS:
Dietary Supplement: Probiotic (VSL#3) — Each subject provided morning stool and venous blood ubes) specimens at three time-points, i.e. at baseline (before probiotic administration), after probiotic administration (VSL#3®, one capsule twice a day) for 4 weeks, and at 4 weeks after stopping the probiotic intake. Each capsule contained approximately 112.5 billion live freeze-dried bacteria (a mixture of eight species -- Streptococcus thermophilus, Bifidobacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, and Lactobacillus delbrueckii), which had been stored at 2-4ºC till ingestion.

SUMMARY:
Healthy human gut contains a large number of bacteria, which belong to several different species. Some genes in these bacteria encode enzymes that the human body cannot produce. These enzymes can catalyze metabolic reactions in the distal small bowel. For instance, bacterial enzymes can breakdown indigestible dietary constituents, making available extra energy to the host. The current paradigm treats the human body as a 'metagenome', i.e. a composite of Homo sapiens genes and genes in the genomes of the colonizing bacteria.

Till recently, accurate determination of bacterial gut flora was not possible. Recent development of multi-parallel sequencing techniques has allowed unbiased determination of profile of gut flora. These techniques have revealed changes in gut flora in several disease conditions, including those of the gastrointestinal tract and liver. This has prompted the use of drugs, such as probiotics to restore the gut flora.

Probiotics contain living microorganisms, and are administered in an attempt to obtain health benefits by restoring normal gut flora. These preparations provide benefit to patients with several diseases, including childhood diarrhea, antibiotic-associated diarrhea, inflammatory bowel disease, vaginitis, etc. However, the mechanisms of their beneficial effects remains unclear. Gut microbiota appear to modulate the development of immune system and maintain a balance between Th17 and T regulatory cells in animals. However, it is not known whether administration of probiotics changes the profile (nature and relative density of various species) of gut flora, and whether these changes are short-lasted or persistent.

This proposal aimed to study whether probiotic administration influences the gut bacterial profile and host immune responses. In addition, we wished to determine whether the changes in gut flora and immune responses persist after probiotic administration is stopped.

DETAILED DESCRIPTION:
Study Subjects The study included 14 healthy non-pregnant women. All subjects provided a written informed consent. The subjects had to (i) be free of systemic (diabetes, autoimmune disease, cancer), gastrointestinal or liver diseases that are known to be associated with alterations in intestinal flora, (ii) be non-obese (body mass index in the range of 20 to 25 Kg/m2), and (iii) not have taken any anti-microbial agent, probiotics, gastric acid suppressant drugs or drugs that alter gastrointestinal motility, in the previous 6 weeks.

Study design Each subject was studied at 3 time points: (i) baseline (enrolment), (ii) after administration of a probiotic in usual dose for four weeks, and (iii) four weeks after discontinuation of probiotic administration. Each subject received Cap VSL#3, 2 capsules daily (each capsule contains 112.5 billion bacteria -- a mixture of 8 bacteria -- Streptococcus thermophilus, Bifido-bacterium breve, Bifidobacterium longum, Bifidobacterium infantis, Lactobacillus acidophilus, Lactobacillus plantarum, Lactobacillus paracasei, and Lactobacillus delbrueckii). At each time point, gut microbiota profile and immune responses were studied.

Metagenomic study for analysis of gut flora Analysis for identification and profiling of gut microflora was done using sequencing of V3 region of the 16S ribosomal ribonucleic acid gene. This gene contains nine variable regions ﬂanked by conserved stretches in all bacteria. Amplification and sequencing of any hypervariable region using specific primers can be used to determine the nature of the bacterium (phylum, family, genus, species, etc). The most widely used regions are V3, V4 and V6; we used V3 region, due to its higher taxonomic resolution.

Stool specimen were collected from subjects at 3 time points as indicated above by asking the subject to pass stool into a clean sterile receptacle; the receptacle was immediately frozen and transported to the laboratory. DNA was isolated from each specimen using standard protocols, quantified, normalised and stored frozen until further use.

Polymerase chain reaction amplification of V3 region was done. Gel-purified amplicons (with different adapter sequences so that data for each sample can be separated at analysis stage) were quantified, normalised and pooled in equimolar quantities (multiplexing). The multiplexed library was subjected to quality control using an Agilent Bioanalyser DNA Chip.

The sequencing library containing V3 amplicons from an equi-amount mixture of various clinical samples was sequenced using an Illumina machine in both directions. The sequence reads were binned according to index sequences, subjected to quality control and sequences in the two directions were fused together to obtain a single read. The sequence data were analysed to determine the profile of gut flora.

Immunological studies Collection of blood specimens Venous blood (6 ml) was collected in lithium heparin/EDTA, at (i) baseline (before starting probiotic administration), (ii) at the end of probiotic treatment (at 4 weeks), and (iii) at 4 weeks after discontinuation of probiotic intake. From 2.5 ml of blood, plasma was separated and stored at -70 degree centigrade. The remaining heparinized blood was used for whole blood culture and for measurement of frequencies of Th17 and Treg cells.

Heparinized blood was used and anti-CD28 (1 ug/ml) for stimulation of T cells and lipopolysaccharide for stimulation of macrophages, in separate wells. Culture supernatants were harvested after 72 hours and stored at -70 degree centigrade. Levels of cytokines (TNF-alpha, IL-10, IFN-gamma, IL-12p70, IL-6 and IL-4) were measured in culture supernatant and plasma using sandwich ELISAs.

Th1, Th2 and Th17 frequencies were determined by stimulation of whole blood with PMA and ionomycin, followed by staining of cells for CD4 and intracellular IFN, IL-4 and IL-1L-17. For Treg enumeration, dual staining for CD4 and Fox-P3 was done.

Ethics considerations The study involves administration of probiotics to healthy subjects. However, these contain bacteria that are a part of the normal gut flora in healthy persons and hence free of any adverse events. In fact, several healthy persons consume these as 'health supplements'. Hence, the administration of these agents should not carry more than minimal risk. The only specimens proposed to be collected are stool specimens and small volumes of blood. No clinical outcomes was collected.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-pregnant women

Exclusion Criteria:

(i) a systemic (diabetes, autoimmune disease, cancer), gastrointestinal or liver disease that is known to be associated with alteration in intestinal microbiota, (ii) obesity or malnutrition (body mass index of <18.5 or >25 Kg/m2), (iii) history of taking an anti-microbial agent, probiotic, or a drug that suppresses gastric acid or alters gastrointestinal motility, in the previous 6 weeks, (iv) any inter-current illness in the last 8 weeks, or (v) a recent change in dietary or bowel habits

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study was planned to study in women only
Enrollment: 14 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Profile of gut flora among healthy Indian women | Baseline
  To determine the profile of gut flora (% abundance of various bacterial phyla, families, genera and species) in healthy Indian women, using a metagenomic technique (sequencing of V3 region of 16S ribosomal RNA).
Effect of probiotic preparation on gut-flora profile | 4 weeks of probiotics administration
  To determine the effect of administration of a probiotic preparation for a 4-week period on the profile of gut flora in healthy Indian women.
Effect of probiotic on immune responses | 4 weeks of probiotics administration
  To assess the effect of probiotic administration on immune responses, and the persistence of such changes on discontinuation of probiotic administration

SECONDARY OUTCOMES:
Persistence of changes, if any, in gut flora after probiotic discontinuation | 4 weeks of discontinuation of probiotics administration
  To determine whether the changes in gut flora after probiotic administration persist after discontinuation of such administration (at 4 weeks after such discontinuation)

IPD SHARING:
Plan to Share IPD: No
We do not have any such plan

REFERENCES:
- [Derived] Singh A, Sarangi AN, Goel A, Srivastava R, Bhargava R, Gaur P, Aggarwal A, Aggarwal R. Effect of administration of a probiotic preparation on gut microbiota and immune response in healthy women in India: an open-label, single-arm pilot study. BMC Gastroenterol. 2018 Jun 15;18(1):85. doi: 10.1186/s12876-018-0819-6. PMID 29907093